CLINICAL TRIAL: NCT07328607
Title: Open Versus Laparoscopic Pancreaticoduodenectomy: A Randomized Controlled Trial
Brief Title: Outcomes After Laparoscopic Versus Open Pancreaticoduodenectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1838/12/2025
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Ampullary Carcinoma; Distal Cholangiocarcinoma; Duodenal Adenocarcinoma; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Pancreaticoduodenectomy (OPD) (Active Comparator): Patients randomized to receive standard open pancreaticoduodenectomy through a bilateral subcostal incision.
  Interventions: Procedure: Open Pancreaticoduodenectomy
- Laparoscopic Pancreaticoduodenectomy (LPD) (Experimental): Patients randomized to receive total laparoscopic pancreaticoduodenectomy using a standardized six-port technique.
  Interventions: Procedure: Laparoscopic Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Open Pancreaticoduodenectomy — Open Pancreaticoduodenectomy with lymphadenectomy and reconstruction via open technique.
  Arms: Open Pancreaticoduodenectomy (OPD)
Procedure: Laparoscopic Pancreaticoduodenectomy — Minimally invasive Whipple procedure using 6 trocars, with specimen extraction via Pfannenstiel incision.
  Arms: Laparoscopic Pancreaticoduodenectomy (LPD)

SUMMARY:
This is a monocentric, prospective, randomized controlled trial comparing the safety and efficacy of laparoscopic pancreaticoduodenectomy (LPD) versus open pancreaticoduodenectomy (OPD). The study aims to determine the morbimortality of the laparoscopic approach compared to the gold standard open approach in adult patients with pancreatic or periampullary lesions.

DETAILED DESCRIPTION:
This is a monocentric, prospective, randomized controlled trial comparing the safety and efficacy of laparoscopic pancreaticoduodenectomy (LPD) versus open pancreaticoduodenectomy (OPD). The study aims to determine the morbimortality of the laparoscopic approach compared to the gold standard open approach in adult patients with pancreatic or periampullary lesions.

This study will randomize 90 eligible patients to receive either LPD or OPD. The primary objective is to compare overall morbidity using the Clavien-Dindo Classification at 90 days postoperative. Secondary objectives include assessment of oncologic outcomes (lymph node harvest, margin status), perioperative metrics (operative time, blood loss), and postoperative recovery (length of stay, readmissions). The study utilizes a prospectively maintained database and adheres to CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed or clinically suspected lesions of: Pancreatic head adenocarcinoma, Ampullary carcinoma, Distal cholangiocarcinoma, Duodenal adenocarcinoma, Pancreatic neuroendocrine tumors, or Intraductal Papillary Mucinous Neoplasm(IPMN) .
* Resectable disease based on preoperative imaging.
* Eastern Cooperative Oncology Group(ECOG) performance status 0-2.
* American Society of Anesthesiologists(ASA )classification I-III.
* Patients able to provide informed consent.

Exclusion Criteria:

* Emergency surgery.
* Previous pancreatic surgery.
* Concurrent major abdominal procedures .
* ASA classification IV or higher.
* Metastatic disease identified preoperatively.
* Locally advanced unresectable disease.
* Active infection or sepsis at time of surgery.
* Severe cardiopulmonary comorbidities precluding major surgery.
* Pregnancy.
* Procedures requiring Total Pancreatectomy, Distal Pancreatectomy, or Enucleation .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Overall Morbidity (Clavien-Dindo Classification) | 90 days postoperative.
  Assessment of all surgical complications graded by severity using the Clavien-Dindo Classification (Grades I-V). Major complications are defined as Grade III or higher.

SECONDARY OUTCOMES:
Number of Lymph Nodes Retrieved | 14 days postoperative.
  Total count of lymph nodes harvested and examined by pathology.
Resection Margin Status (R0/R1/R2) | 14 days postoperative.
  Pathological assessment of margins (Pancreatic neck, bile duct, retroperitoneal, etc.) classified as R0 (>1mm), R1 (≤1mm), or R2 (macroscopic).
Operative Time | Intraoperative
  Time measured from skin incision to skin closure.
Estimated Blood Loss | Intraoperative
  Total blood loss recorded by the anesthesiology team.
Length of Hospital Stay | Up to 90 days.
  Total number of days from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adam MA, Choudhury K, Dinan MA, Reed SD, Scheri RP, Blazer DG 3rd, Roman SA, Sosa JA. Minimally Invasive Versus Open Pancreaticoduodenectomy for Cancer: Practice Patterns and Short-term Outcomes Among 7061 Patients. Ann Surg. 2015 Aug;262(2):372-7. doi: 10.1097/SLA.0000000000001055. PMID 26158612
- [Result] Poves I, Burdio F, Morato O, Iglesias M, Radosevic A, Ilzarbe L, Visa L, Grande L. Comparison of Perioperative Outcomes Between Laparoscopic and Open Approach for Pancreatoduodenectomy: The PADULAP Randomized Controlled Trial. Ann Surg. 2018 Nov;268(5):731-739. doi: 10.1097/SLA.0000000000002893. PMID 30138162